CLINICAL TRIAL: NCT01870973
Title: Effect on Initial Endodontic Treatment on Postoperative Pain in Symptomatic Teeth With Pulpal Necrosis
Brief Title: Effect of Root Canal Treatment (Versus no Treatment) for Patients With Tooth Infections and Toothaches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Melissa Drum, Associate Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: root canal versus no treatment
Record Dates: First submitted 2013-06-04; First posted 2013-06-06 (Estimated); Results first posted 2015-06-18 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-06

CONDITIONS: Postoperative Pain
Keywords: postoperative pain; root canal treatment
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia; Anti-Bacterial Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- root canal treatment (Experimental): root canal treatment, anesthesia with 2% lidocaine with 1:100,000 epinephrine, pain medication (1000 mg acetaminophen and 600 mg ibuprofen every 6 hours)five day supply, antibiotic (500 mg penicillin, if allergic 300 mg clindamycin)
  Interventions: Procedure: root canal treatment, anesthesia, pain medications, and antibiotic
- no root canal treatment (Active Comparator): no root canal treatment, anesthesia with 2% lidocaine with 1:100,000 epinephrine, pain medication (1000 mg acetaminophen and 600 mg ibuprofen every 6 hours)five day supply, antibiotic (500 mg penicillin if allergic 300 mg clindamycin)
  Interventions: Procedure: no root canal treatment, anesthesia, pain medications, and antibiotic

INTERVENTIONS:
Procedure: root canal treatment, anesthesia, pain medications, and antibiotic — Root canal treatment is the intervention (no initial treatment versus initial treatment). We are not studying a drug or device.
  Arms: root canal treatment
Procedure: no root canal treatment, anesthesia, pain medications, and antibiotic
  Arms: no root canal treatment

SUMMARY:
The purpose of this study is to evaluate patients with emergency pain and a sore (infected) tooth to determine if immediate root canal therapy is better at reducing pain, when compared to initial treatment with antibiotic and pain medication followed by root canal therapy. Each participant will be randomly assigned a number, which will determine if they will receive initial endodontic treatment that day or at a later date. Each participant will receive an anesthetic injection, pain medication and a prescription for an antibiotic. They will be asked to keep a diary to record their pain level after the injection and their pain levels and the amount and type of pain medication taken each day for the next 5 days. Participants who did not receive root canal therapy at the initial appointment will receive it after the 5 day postoperative period. The pain levels and medication use will be compared between the treatment and nontreatment groups.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* in good health (ASA classification I or II)
* able to give informed consent
* infected tooth with toothache (symptomatic tooth with pulpal necrosis)

Exclusion Criteria:

* allergy to ibuprofen, acetaminophen or codeine
* history of significant medical problems (ASA classification III or greater)
* angioedema or bronchospastic reactivity to aspirin or other NSAIDs
* pregnant or lactating
* inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2013-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University College of Dentistry, Postle Hall, Columbus, Ohio, United States

REFERENCES:
- [Background] Houck V, Reader A, Beck M, Nist R, Weaver J. Effect of trephination on postoperative pain and swelling in symptomatic necrotic teeth. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2000 Oct;90(4):507-13. doi: 10.1067/moe.2000.108960. PMID 11027389
- [Background] Nist E, Reader A, Beck M. Effect of apical trephination on postoperative pain and swelling in symptomatic necrotic teeth. J Endod. 2001 Jun;27(6):415-20. doi: 10.1097/00004770-200106000-00013. PMID 11487138
- [Background] Henry M, Reader A, Beck M. Effect of penicillin on postoperative endodontic pain and swelling in symptomatic necrotic teeth. J Endod. 2001 Feb;27(2):117-23. doi: 10.1097/00004770-200102000-00016. PMID 11491635
- [Background] Nusstein JM, Reader A, Beck M. Effect of drainage upon access on postoperative endodontic pain and swelling in symptomatic necrotic teeth. J Endod. 2002 Aug;28(8):584-8. doi: 10.1097/00004770-200208000-00005. PMID 12184419
- [Background] Mickel AK, Wright AP, Chogle S, Jones JJ, Kantorovich I, Curd F. An analysis of current analgesic preferences for endodontic pain management. J Endod. 2006 Dec;32(12):1146-54. doi: 10.1016/j.joen.2006.07.015. Epub 2006 Oct 19. PMID 17174670
- [Background] Wells LK, Drum M, Nusstein J, Reader A, Beck M. Efficacy of Ibuprofen and ibuprofen/acetaminophen on postoperative pain in symptomatic patients with a pulpal diagnosis of necrosis. J Endod. 2011 Dec;37(12):1608-12. doi: 10.1016/j.joen.2011.08.026. Epub 2011 Oct 1. PMID 22099891

RESULTS

PARTICIPANT FLOW:
Groups:
- Root Canal Treatment: root canal treatment, anesthesia with 2% lidocaine with 1:100,000 epinephrine, pain medication (1000 mg acetaminophen and 600 mg ibuprofen every 6 hours)five day supply, antibiotic (500 mg penicillin, if allergic 300 mg clindamycin)
  root canal treatment: Root canal treatment is the intervention (no initial treatment versus initial treatment). We are not studying a drug or device.
- no Root Canal Treatment: no root canal treatment, anesthesia with 2% lidocaine with 1:100,000 epinephrine, pain medication (1000 mg acetaminophen and 600 mg ibuprofen every 6 hours)five day supply, antibiotic (500 mg penicillin if allergic 300 mg clindamycin)
  no root canal treatment
Period: Overall Study
Arm/Group | Root Canal Treatment | no Root Canal Treatment
Started | 56 | 52
Completed | 46 | 49
Not Completed | 10 | 3
Not completed — Lost to Follow-up | 10 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Root Canal Treatment | no Root Canal Treatment | Total
Number analyzed (Participants) | 46 | 49 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.3 (12.1) | 39.1 (16.1) | 37.7 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 25 | 45
  Male | 26 | 24 | 50
Region of Enrollment [Number; unit: participants]
  United States | 46 | 49 | 95

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients With Success as Defined by no or Mild Pain as Analyzed on a VAS Scale and no Narcotic Use
Description: pain measurement as assessed on a visual analog scale and pain medication usage
  definition of success = no or mild pain as analyzed on VAS scale and no narcotic use; analyzed by logistic regression
  VAS scale is 0 to 170 mm with the higher numbers indicating more pain and less success.
Time Frame: each day for 5 days
Measure: Number; unit: percentage of participants
Arm/Group | Root Canal Treatment | no Root Canal Treatment
Number analyzed (Participants) | 46 | 49
percentage of participants | 52 | 43

ADVERSE EVENTS:
Arm/Group | Root Canal Treatment | no Root Canal Treatment
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/52
Other Adverse Events (participants affected / at risk) | 0/56 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No